CLINICAL TRIAL: NCT01576003
Title: Efficacy of Enteral Glutamine in Reducing Bloodstream Infections in Short Bowel Syndrome Infants
Brief Title: Enteral Glutamine in Reducing Bloodstream Infections in Short Bowel Syndrome Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Emmaus Medical, Inc. (Industry); University of Michigan (Other); Emory University (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-2706; 1R21DK088027-01A1 (NIH)
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Bloodstream Infections; Short Bowel Syndrome; Development; Nutrition; Biological Markers
Keywords: Short Bowel Syndrome; Necrotizing Entercolitis (NEC); Atresia; Parenteral Nutrition; Biological Markers; Growth
MeSH Terms: conditions — Sepsis; Short Bowel Syndrome; Hyperphagia | interventions — Glutamine; Alanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Glutamine (Experimental): Infants randomized to the Glutamine group will receive L-Glutamine (GLN) administered enterally at a dose of 0.6g/kg body weight/day (0.3g/kg/dose) in 2 divided daily doses for 6 months. GLN will be dissolved in water, breast milk or formula and administered to the subject orally or through their enterostomy tube approximately every 12 hours (twice a day).
  Interventions: Drug: Glutamine
- L-alanine (Placebo Comparator): Infants randomized to the placebo group will receive L-alanine (ALA) administered enterally at a dose of 0.6g/kg body weight/day in 2 divided doses (0.3g/kg/day twice a day) for 6 months. ALA will be dissolved in water, breast milk or formula and administered to the subject orally or through their enterostomy tube approximately every 12 hours (twice a day).
  Interventions: Dietary Supplement: L-alanine
- Healthy Control (No Intervention): Healthy age-matched infants (n=12) will have serial stools collected on 4 occasions, each separated by 60 days.

INTERVENTIONS:
Drug: Glutamine — 0.3 g/kg, taken orally/feeding tube every 12 hours/twice a day for 180 days (6 months)
  Other Names: NutreStore
  Arms: Glutamine
Dietary Supplement: L-alanine — 0.3 g/kg, taken orally/feeding tube every 12 hours/twice a day for 180 day (6 months)
  Arms: L-alanine

SUMMARY:
The purpose of this research study is to evaluate the effects (good and bad) of supplementation with Glutamine to that of a placebo (L-alanine), on your child and their Short Bowel Syndrome. Researchers are doing this study to see if the addition of Glutamine to oral/tube feeding (nutrition therapy) will work better by preventing bloodstream infections, improving growth, and/or changing the make-up of bacteria in your child's intestine. Glutamine is approved by the FDA for use in adults with Short Bowel Syndrome. In this study, the investigators will be assessing how well Glutamine affects Short Bowel Syndrome in children.

DETAILED DESCRIPTION:
This is a double-blind, randomized placebo-controlled pilot study to investigate the efficacy of enteral glutamine (GLN) supplementation in 36 infants, ≤ 12 months of age with parenteral nutrition (PN)-dependent short bowel syndrome (SBS) due to massive small bowel resection for NEC and/or atresia on improving weaning of PN and preventing infections. The investigators intend to evaluate the effect of enteral feeding and GLN supplementation on the gut bacteria. The investigators will also recruit 12 age-matched controls to evaluate the normal gut bacteria.

ELIGIBILITY:
Inclusion Criteria for Controls:

* Less than or equal to 12 months of age
* Normal small bowel length without any intestinal resection or primary intestinal disease
* Not currently on Total Parenteral Nutrition (TPN) and if ever on TPN this should have been discontinued for at least 4 weeks.

Exclusion Criteria for Controls:

* Major congenital or chromosomal anomalies
* Inability to tolerate enteral nutrition/regular cow's milk, breast milk or formula
* History of liver/intestinal transplantation

Inclusion Criteria for Glutamine and Placebo Group of Short Bowel Syndrome (SBS) Patients:

* Less than or equal to 12 months of age
* Patients who have undergone small bowel resection due to necrotizing enterocolitis (NEC) or intestinal atresia with known small bowel length
* Patients who have been Parenteral Nutrition (PN) dependent for more than 42 consecutive days and currently on TPN at time of enrollment
* Patients who have the ability to take partial enteral nutrition or breast milk or elemental formula to allow the appropriate dose of glutamine or placebo
* Signed informed consent for the use of Glutamine or placebo

Exclusion Criteria for Glutamine and Placebo Group of SBS Patients:

* Major congenital or chromosomal anomalies
* Inability to tolerate enteral nutrition that will preclude treatment with enteral Glutamine or L-alanine placebo for > 2 weeks
* Liver/Intestinal transplantation

Ages: 6 Weeks to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2012-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Conrad R Cole, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - C.S. Mott Children's Hosptial, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant consented and then withdrew prior completing any study procedure. This participant is not included in the participant flow due to the fact no study procedures or randomization occurred.
Groups:
- Glutamine: L-Glutamine: 0.3 g/kg, taken orally/feeding tube every 12 hours/twice a day for 180 days (6 months)
- Placebo: L-alanine: 0.3 g/kg, taken orally/feeding tube every 12 hours/twice a day for 180 day (6 months)
- Healthy Control: No Intervention - Healthy age-matched infants provided stools on 4 occasions, each separated by 60 days.
Period: Overall Study
Arm/Group | Glutamine | Placebo | Healthy Control
Started | 2 | 3 | 4
Completed | 1 | 1 | 4
Not Completed | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: 1 Participant withdrew in the screening phase and did not randomize.
Groups:
- Placebo: L-Alanine: 0.3 g/kg, taken orally/feeding tube every 12 hours/twice a day for 180 days (6 months)
- Total: Total of all reporting groups
Arm/Group | Glutamine | Placebo | Healthy Control | Total
Number analyzed (Participants) | 2 | 3 | 4 | 9
Age, Customized [Count of Participants; unit: Participants]
  6 weeks through 2 months | 0 | 0 | 1 | 1
  3 months through 4 months | 0 | 1 | 1 | 2
  5 months through 6 months | 1 | 0 | 1 | 2
  7 months through 8 months | 1 | 0 | 1 | 2
  9 months through 10 months | 0 | 2 | 0 | 2
  11 months through 12 months | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 3
  Male | 1 | 1 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Cause of Short Bowel Resection [Count of Participants; unit: Participants]
  Atresia | 1 | 1 | 0 | 2
  Necrotizing enterocolitis (NEC) | 1 | 0 | 0 | 1
  NEC and Atresia | 0 | 2 | 0 | 2
Birth Weight [Mean (Full Range); unit: kilograms] — Population: Birth weight data was not obtained on healthy controls.
  kilograms
    number analyzed (Participants) | 2 | 3 | 0 | 5
    (all) | 2.4 [1.85 to 2.9] | 2.6 [2.3 to 2.9] |  | 2.35 [1.85 to 2.9]
Bowel Length [Mean (Full Range); unit: Centimeters] — Population: Healthy Controls did not have a bowel resection.
  Centimeters
    number analyzed (Participants) | 2 | 3 | 0 | 5
    (all) | 49.5 [33.0 to 66.0] | 82.0 [45.0 to 150.0] |  | 69.0 [33.0 to 150]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Bloodstream Infections (BSI)
Description: Evaluate the efficacy of enteral Glutamine supplementation to decrease bloodstream infections in participants that are parenteral nutrition dependent with Short Bowel Syndrome due to necrotizing enterocolitis (NEC) and/or atresia.
Time Frame: 6 months
Population: Two of the five participants analyzed completed the study. Healthy controls did not receive parenteral nutrition and were not analyzed in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Glutamine | Placebo
Number analyzed (Participants) | 2 | 3
Participants | 0 | 1

2. Primary Outcome: Length Velocity
Description: Assess the efficacy of 6 months of therapy with enteral Glutamine on length velocity.
Time Frame: 6 months
Population: The number analyzed at Baseline and days 60, 120 and 180 differ from the overall number analyzed due protocol noncompliance and participant request to withdrawal from the protocol. Healthy controls were not analyzed in this outcome measure because they did not receive parenteral nutrition, L-Glutamine or placebo.
Measure: Mean (Full Range); unit: Centimeters
Arm/Group | Glutamine | Placebo
Number analyzed (Participants) | 2 | 3
Centimeters
  Length at Baseline | 60.9 [56.7 to 65.0] | 66.0 [63.2 to 70.8]
  Length at Day 60: number analyzed (Participants) | 1 | 3
  Length at Day 60 | 62.2 | 67.5 [63.6 to 71.4]
  Length at Day 120: number analyzed (Participants) | 1 | 1
  Length at Day 120 | 66.8 | 73.7
  Length at Day 180: number analyzed (Participants) | 1 | 1
  Length at Day 180 | 68 | 78.2

3. Secondary Outcome: Head Circumference
Description: Assess the efficacy of 6 months of therapy with enteral Glutamine on head circumference
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Full Range); unit: Centimeters
Arm/Group | Glutamine | Placebo
Number analyzed (Participants) | 2 | 3
Centimeters
  Head Circumference at Baseline | 42.9 [41.1 to 44.8] | 43.8 [42.2 to 46.8]
  Head Circumference at Day 60: number analyzed (Participants) | 1 | 3
  Head Circumference at Day 60 | 43.5 | 43.4 [42.0 to 44.8]
  Head Circumference at Day 120: number analyzed (Participants) | 1 | 1
  Head Circumference at Day 120 | 48.8 | 46
  Head Circumference at day 180: number analyzed (Participants) | 1 | 1
  Head Circumference at day 180 | 44.5 | 46.6

4. Secondary Outcome: Mid Arm Circumference
Description: Assess the efficacy of 6 months of therapy with enteral Glutamine on mid arm circumference.
Time Frame: 6 months
Population: The number analyzed at Baseline and days 60,120 and 180 differ from the overall number analyzed due protocol noncompliance and participant request to withdrawal from the protocol. Healthy controls were not analyzed in this outcome measure because they did not receive parenteral nutrition, L-Glutamine or placebo.
Measure: Mean (Full Range); unit: Centimeters
Arm/Group | Glutamine | Placebo
Number analyzed (Participants) | 2 | 3
Centimeters
  Mid Arm Circumference at Baseline | 13 [10.9 to 15.0] | 16.0 [16.0 to 16.0]
  Mid Arm Circumference at Day 60: number analyzed (Participants) | 1 | 3
  Mid Arm Circumference at Day 60 | 12.6 | 16.0 [15.8 to 16.3]
  Mid Arm Circumference at Day 120: number analyzed (Participants) | 1 | 1
  Mid Arm Circumference at Day 120 | 12.5 | 8.8
  Mid Arm Circumference at day 180: number analyzed (Participants) | 1 | 1
  Mid Arm Circumference at day 180 | 12.8 | 17.3

5. Secondary Outcome: Weight Velocity
Description: Assess the efficacy of 6 months of therapy with enteral Glutamine on weight velocity.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Full Range); unit: Kilograms
Arm/Group | Glutamine | Placebo
Number analyzed (Participants) | 2 | 3
Kilograms
  Weight at Baseline | 6.5 [5.2 to 7.9] | 8.1 [7.6 to 9.2]
  Weight at Day 60: number analyzed (Participants) | 1 | 3
  Weight at Day 60 | 6.4 | 8.4 [7.8 to 9.0]
  Weight at Day 120: number analyzed (Participants) | 1 | 1
  Weight at Day 120 | 7.1 | 9.3
  Weight at day 180: number analyzed (Participants) | 1 | 1
  Weight at day 180 | 7.9 | 9.4

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Glutamine | Placebo | Healthy Control
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/3 | 0/4
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glutamine (N=2) | Placebo (N=3) | Healthy Control (N=4)
Viral Illness (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hospitalization for fever in a patient with a central line (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Respiratory syncytial virus (RSV) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glutamine (N=2) | Placebo (N=3) | Healthy Control (N=4)
Diaper Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Otitis Media (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (General disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Central Venous Catheter (CVC) dislodged (General disorders) | 1 (1) | 0 (0) | 0 (0)
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Recruitment was low due to the improvement in care from the use of ethanol lock therapy and improved techniques related to line care. Early termination of participants lead to small number of subjects analyzed and inability to analyze all study aims.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT01576003/Prot_SAP_000.pdf